CLINICAL TRIAL: NCT07237971
Title: Cocreating Action to Improve Rationality in the Health System
Acronym: CAIR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Lucy Anne Parker, Associate professor, Universidad Miguel Hernandez de Elche
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Grant No. 101125843; ERC-2023-COG 101125843 (Other Grant/Funding Number: European Research Council (ERC) through the Horizon Europe Framework Programme for Research and Innovation)
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Health-Related Quality-of-Life; Social Capital; Health Literacy; Community Based Participatory Research; Antibiotic Prescription; Mental Health Literacy; Cardio Vascular Disease; Antimicrobial Drug Resistance; Well-being; Health Equity
Keywords: Community health; Cocreation action; Health system; Health literacy; Social capital; Community capital; Antibiotic drug use; Cardiovascular drug use; Psychotropic drug use; Health-related quality of life; Health equity
MeSH Terms: interventions — Community-Based Participatory Research

STUDY DESIGN:
Intervention Model Description: A community-based participatory research will be conducted to engage citizen scientists in the cocreation of community-led actions to promote psychological well-being, CV health, and prevent antimicrobial resistance. The design, implementation, and evaluation of the actions will apply an assets-based approach in an iterative manner over 3 years. The investigators will use some preliminary results from a population survey, a survey of patients collecting their medication at community pharmacies, aggregate health service indicators on medication consumption and primary care consultations, and qualitative methods (sociograms, interviews, and focus groups) to boost the cocreation process. Finally, the impact of the cocreated actions will analysed. This study will use a before-after comparison of survey indicators, an interrupted time-series analysis of health service data and qualitative analysis.
Masking Description: No parties are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cocreating process to improve rationality in the health system in a deprived neighborhood (Experimental)
  Interventions: Other: Cocreation process

INTERVENTIONS:
Other: Cocreation process — The cocreation process will involve various advisory and participatory bodies to ensure the active involvement of the community and local institutions, also with the research team, ensuring that actions respond to collective needs of the community. Recruitment of these advisory and participatory bodies will be carried out through a participatory strategy involving the Basic Health Councils of the healthcare centers in the area, as well as other associations, religious institutions, and local leaders. Based on previous sociograms, strategic locations will be identified for organizing informational meetings in accessible places in the area, such as community centers. Dissemination will be carried out through social media, posters, and other inclusive means to ensure the participation of vulnerable groups. Participation in the cocreation process will be open, voluntary, and will depend on the interest of individuals and entities in the area.
  Other Names: Community-based participatory research (CBPR)

SUMMARY:
Despite widespread recognition of social, economic, or environmental health determinants, health action remains heavily dominated by individual-level solutions (e.g., medication, patient counselling, vaccination). This study aims to stimulate changes in health system functioning by demonstrating how the cocreation of actions to address psychological well-being, cardiovascular health, and antimicrobial resistance from within the community can alleviate the burden on primary care services, reduce medicalisation and increase health equity.

The scientific approach uses mixed methods and incorporates theory from multiple disciplines. This study will appraise how the current system addresses psychological well-being, cardiovascular (CV) health, and rational use of antibiotics using a population survey, a survey of patients collecting their medication at community pharmacies, aggregate health service indicators on medication consumption and primary care consultations, and qualitative methods exploring stakeholders' perceptions.The investigators will undertake community-based participatory research to engage citizen scientists in the cocreation of community-led actions to promote psychological well-being, CV health, and prevent antimicrobial resistance. The design, implementation, and evaluation of the actions will apply an assets-based approach and apply theories and frameworks from implementation science in an iterative manner over 3 years. Finally, the impact of the cocreated actions will be analysed, considering effectiveness and broader contextual issues such as initiative adoption, implementation, and maintenance. The investigators will use a before-after comparison of survey indicators, an interrupted time-series analysis of health service data and qualitative analysis.

The goal is to demonstrate how the integration of community action with attention to the social determinants of health, can lead to a more rational approach to health care and ultimately improve health and health equity.

DETAILED DESCRIPTION:
This study seeks to cocreate actions that address three major health issues within the community to reduce medicalisation and help unburden primary healthcare services. The first issue is related to psychological well-being and the overuse of anxiolytics and antidepressants. Mental health problems are one of the greatest public health challenges in the European Region, affecting about 25% of the population every year and some estimates place Spain, where this research takes place, as the highest per-capita consumer of anxiolytic medication in the world. The second issue relates to addressing CV health and over-reliance on medication to treat CV risk factors as "pre-diseases". While CV disease continues to be the leading cause of adult mortality worldwide, there is a rise in overdiagnosis and overtreatment of CV risk factors in primary care and limited CV health promotion at community level. The third issue is to promote rational use of antibiotics and reduce the risk of antimicrobial resistance, an issue considered to be in the top 10 global public health threats today.

As the title of this study suggests, the investigators question whether the current approach to these important public health issues is truly rational. Health action remains heavily dominated by individual-level solutions (e.g., medication, patient counselling, vaccination) despite widespread recognition of the social, economic, or environmental factors that determine health. Health professionals frequently acknowledge the importance and potential of non-pharmacological community-based interventions, yet barriers exist to put them into practice. Even the way that the public health system is conceptualised leads to overemphasize the importance of the health services as the accountable component for providing health and well-being. In fact, there are numerous organizations and individuals who develop actions in areas that are not directly recognizable as part of the health system (e.g., senior citizens clubs, urban planners, cultural centres), but which greatly facilitate the effectiveness of the system and have the potential to produce significant health and wellbeing benefits. The project will apply a "systems thinking" approach and consider that any organization, person, or action that influences the physical or social environment has the potential to influence health and wellbeing, and thus could be considered part of the public health system if they are incorporated into the decision-making domains that have a primary desire or interest in maximizing health. Important, yet frequently underestimated, health systems components are found in the community.

Identifying and activating health promoting resources in the community is a legitimate and effective way to improve health and health equity. It forms the basis of a substantial body of research and practice on health promotion with community assets. A community can also be characterised and described by its level of social capital, which in itself is a key component of community resources, as well as a determinant of physical and mental health. It includes the perceptions that people have about the level of interpersonal trust, exchange and reciprocity in their community, as well as the density of their social networks and patterns of civic engagement. This study put forward an ambitious plan to show how the power of the community and its members can be harnessed to cocreate actions that move them from a predominant biomedical vision to a truly rational health system.

Engaging the community in research or practice is acknowledged as a powerful tool to elicit meaningful and sustainable change. Furthermore, it is an effective way to reduce inequity. In this line, increasing attention is centred on developing citizen science initiatives that move beyond engaging citizens in data collection, and towards citizens having a meaningful input in all phases of the research, including design and translation of the findings into practice. The community-based participatory research model has proven useful in this endeavour. This study considers here that deep community engagement in research can improve critical health literacy (CHL), not just among the citizen scientists but among the community as a whole. CHL refers to individuals or communities that are able to critically appraise information, understand the social determinants of health and have skills oriented towards collective social and political action. The issue is paramount to the problem addressed here as CHL is widely assumed to lead to a more effective and efficient use of health services. In light of these considerations, the research proposed seeks to foster the complexity and dynamism of the health system by integrating community action and attention to the social determinants of health. This will refocus how psychological wellbeing, CV health, and antimicrobial resistance are approached. Together with citizen scientists the investigators will cocreate community actions in each of these 3 areas and will show how they can ultimately impact health and health equity. The objectives are:

Overall objective: To determine the impact on health and health equity of a series of cocreated actions to improve rationality in the health system.

Specific objectives:

1. To generate rigorous quantitative and qualitative epidemiological data on the current health systems approach to address psychological wellbeing, CV health, and antimicrobial resistance.
2. To cocreate actions to promote psychological wellbeing, CV health, and rational use of antibiotics with a community approach.
3. To assess the impact of the cocreated actions on health and health equity at local population level.

ELIGIBILITY:
Survey general population:

A representative population survey of adult (aged 18 years and over) who are residents in the Municipal District 2 of Elche (Spain).

Survey community pharmacies:

Individuals who visit the pharmacies collaborating in the Municipal District 2 of Elche (Spain) to obtain any of the medications, aged 18 years and over for three a priori established medication groups.

* Group 1 (Antidepressants and Anxiolytics): N05B, N05C, N06A.
* Group 2 (Cardiovascular disease risk factor medication): A10B (antidiabetics), C10A (cholesterol-lowering drugs), C07A, C09A, C03C, C08C (antihypertensives).
* Group 3 (Antibiotics): J01

Health service data from primary care:

A series of aggregate indicators will be collected from the electronic information systems of the regional health authorities (Conselleria de Sanidad de la Generalitat Valenciana), which hosts information on both prescriptions made by physicians and those dispensed in the community pharmacies of the Valencian Community. These indicators will be calculated for individuals aged 18 years and over for groups 2 and 3, and 12 years and over for group 1 using aggregate data from health system's registries and, therefore, not considering 12 years old as minimum age limit of the eligible participants in the present study protocol registry. Furthermore, aggregate data about the number of consultations will be collected in the two primary care facilities in the study area for individuals aged 18 and over.

Qualitative methods and cocreation procedure:

Focus groups, sociograms and in-depth interviews will include 6-8 participants and last approximately 90 minutes. Participation in the co-creation process will be open, voluntary, and will depend on the interest of individuals and entities in the area. Eligibility criteria:

* People aged 18 and over who are residents or have a job or family connection in the Municipal District 2 of Elche (Spain) who are interested in participating, wish to be actively involved in the co-creation, planning, and implementation of community initiatives, and are available to attend the conferences, meetings, and workshops.
* Representatives from community institutions and associations, including professionals from the Elche Public Health Center, primary care teams in the area, Elche Council staff, as well as professionals and volunteers from NGOs and other local organizations with experience in community work in the district.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 5 years
  Health-related quality of life will be measured using the VR-12 questionnaire, which was internationally validated (Selim et al., 2022). The VR-12 questionnaire contains 12 items that assess eight aspects of health-related quality of life: physical dimension, mental dimension, physical function, physical role, bodily pain, general health, vitality, emotional role, social function, and mental health. The instrument measures eight scales that are used to produce a summary score in two different dimensions: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS).
Medical drug consumption | 5 years
  Aggregated data of Primary Care for the studied Basic Health Zones (BHZ):
  * Defined Daily Dose (DDD) per 1,000 inhabitants per day of drugs in classes N05B, N05C, and N06A prescribed to people over 12 years of age by an SNS professional in each basic health zone (BHZ).
  * DDD of drugs of classes N05B, N05C, and N06A that have been prescribed to persons over 12 years in each BHZ and are subsequently dispensed in a community pharmacy.
  * DDD of drugs of classes A10B, C10A, C07A, C09A, C03C, C08C prescribed to persons over 15 years in each BHZ.
  * DDD of drugs of classes A10B, C10A, C07A, C09A, C03C, C08C that have been prescribed to people over 15 years in each BHZ and are subsequently dispensed in a community pharmacy.
  * DDD of drugs of classes J01 prescribed to people over 15 years in each BHZ.
  * DDD of drugs of classes J01 that have been prescribed in each BHZ and are subsequently dispensed in a community pharmacy.
Workload in primary healthcare | 5 years
  The number of consultations carried out in each studied Basic Health Zone will be retrieved for people over 15 years, disaggregated by the reason for consultation. This indicator will be calculated monthly during the five years of the study and disaggregated by relevant sociodemographic characteristics. Similarly, the average number of medications per clinical encounter will be calculated by dividing the total number of prescriptions in each period by the total number of consultations. Similarly, at six-month intervals, the percentage of clinical encounters that result in the prescription of antibiotics will be computed.

SECONDARY OUTCOMES:
Critical Health literacy | 5 years
  Different domains of health literacy include basic functional health literacy (the ability to access, understand, evaluate, and apply health information), communicative health literacy, and critical health literacy (Nutbeam, 2020). This study is particularly concerned with critical health literacy because it involves the critical evaluation of information, understanding the social determinants of health, and is linked to collective action (Chinn, 2011). Furthermore, it is widely assumed that better critical health literacy leads to more effective and efficient use of services (Sykes et al., 2013). These aspects will be measured using the All Aspects of Health Literacy Scale (Chinn & McCarthy, 2013) after analyzing the psychometric properties of a new version adapted to Spain scoring between 1 (lowest health literacy) and 43 (highest health literacy).
Social capital and community belonging | 5 years
  A measure related to social capital will be included, given that it is a key determinant of physical and mental health (Kawachi et al., 1999; Stoyanova & Díaz-Serrano, 2009; Villalonga-Olives & Kawachi, 2015). This study will develop a questionnaire based on a scale previously validated in the United States for Latino population (Villalonga-Olives et al., 2016). This study will focus on trust in close friends and family to cope with difficult times (e.g., the possibility of receiving financial help in times of need or having someone to care for children in an emergency) and community belonging, also including a domain of social cohesion from the Canadian Community Health Survey. Social capital will score between 0 (lowest social capital) and 10 (highest social capital), social cohesion between 8 (lowest cohesion) and 33 (highest cohesion), and community belonging between 6 (lowest belonging) and 24 (highest belonging).
Community capital | 5 years
  An ad-hoc tool will be developed to measure the use of community assets, here defined as "any factor (or resource) that enhances the capacity of individuals, groups, communities, populations, social systems and institutions to maintain and sustain health and well-being and helps them to reduce health inequalities", as well as potential barriers to their use. The tool will contain questions on community assets, classified into seven categories: 1. Natural, 2. Cultural, 3. Human, 4. Social, 5. Political, 6. Financial and 7. Built. Participants will be asked if they consider that their environment (this includes the neighbourhood where they live, and other places in the municipality that they frequent) has these community assets and how often they use them. The ad-hoc instrument will be pre-tested with a small representative sample of the community to obtain feedback on the clarity and relevance of the questions in order to make any necessary adjustments before its final implementation.
Knowledge, attitudes and practices on personal antibiotic use | 5 years
  Knowledge, attitudes and practices on personal antibiotic use will be measured using an instrument validated in Spain. This instrument will obtain data to analyse common antibiotic-related behaviours of the following three dimensions: knowledge (what respondents know about antibiotics), attitude (what respondents think about antibiotics) and practice (what they do regarding antibiotics). The different domains will be measured in a Likert scale from 0 to 10 with a final score between 0 (lowest knowledge, attitudes and practices on personal antibiotic use) and 160 (highest knowledge, attitudes and practices).
Mental health literacy | 5 years
  The investigators will use the brief mental health literacy questionnaire for adults by Campos et al. (2022). For its validation in Spain, this study will carry out its translation and cultural adaptation through direct translation, expert review, back-translation, and semantic adjustments. This study will then validate its content through consultation with mental health specialists to assess the clarity and relevance of the items. A pilot test will be carried out on a small sample of participants who visit the community pharmacy to detect possible comprehension problems. Moreover, psychometric validation will be carried out with a representative sample, evaluating internal consistency (Cronbach's alpha), construct validity (factor analysis), and test-retest reliability. Mental health literacy will be measured using a Likert scale from 1 to 5, with a final score between 16 (lowest mental health literacy) and 80 (highest mental health literacy).
Use and barriers to non-pharmacological interventions | 5 years
  The investigators will present a list of non-pharmacological interventions for the patients to select if some of them have been offered by their clinicians, family members, friends or other means. Furthermore they will report on perceived barriers to following non-pharmacological interventions. The questionnaire tool will be developed and validated.
Knowledge about behaviours and cardiovascular risk | 5 years
  The level of knowledge and attitude toward behaviours related to CV health and risk will be assessed using the questionnaire validated in Spain. The questionnaire is scored using a 5-point Likert scale, where 1 represents the least correct answer and 5 the most correct, with a minimum score of 24 (lowest level of knowledge) maximum score of 120 (highest level of knowledge) points for the 24 items. A score above 90 indicates a high level of knowledge (at least 75% correct answers).
Antibiotic appropriateness | 5 years
  To assess antibiotic appropriateness, we will use the TARGET antibiotic checklist, included in the TARGET antibiotic toolkit ("treating antibiotics responsibly; guidance, education and tools") developed by the UK Royal College of General Practitioners in 2022.
Medication knowledge | 5 years
  Patients' knowledge of their medications will be assessed, including aspects such as indication, duration of treatment, method of administration, and possible adverse effects, using a questionnaire validated in Spain. This questionnaire will be applied to a single medication per participant in the pharmacy survey. It is assumed that in a more rational healthcare system, people take fewer medications as a more appropriate and justified use of treatments. At the same time, those who do need medication may have greater knowledge about it, given that in a more efficient system there is better health literacy and patients have more time with their healthcare professional to receive detailed explanations about their treatment.
Indicators of the National Antibiotic Resistance Plan | 5 years
  The Spanish National Antibiotic Resistance Plan includes a selection of indicators for analysing antimicrobial consumption in primary care. These indicators are designed to measure both consumption rates and exposure to antibiotics among the population and to analyse the selection of certain groups of antibiotics.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Community, Elche, Alicante
  - Community based. Municipal District 2 of Elche, Elche, Alicante

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated by the CAIR project will be archived in the data repository Zenodo and will be linked on the project's website https://www.cairproject.eu/.
  Metadata from Zenodo (title, description, keywords, creation date, creators, license, and format) will be used for dataset description and discovery.
  DOIs will be assigned to datasets published in this repository to ensure unique citation, while Zenodo will provide secure storage for our (meta)data and allow us different licenses and access levels.
  The DOI of (meta)data will be included in relevant publications, making it easy to locate the anonymized raw data.
  The more public-facing content will also be disseminated through the project's associated social media channels as Facebook (CAIR Project), Bluesky (@erc.europa.eu), and Instagram (cairproject.eu)).
Supporting Information: Study Protocol
Time Frame: From October 2025 to April 2029
Access Criteria: The Creative Commons Attribution 4.0 International (CC BY 4.0) license will be used for our anonymized data, which will be stored on Zenodo. This license allows others to use, reproduce and disseminate out data (free of charge for any user). Data will remain available indefinitely, but it will need researchers' permission by a written request. Any use of data should always include proper attribution and not modify the content.
  Any embargo will not be applied on the open data; however, an embargo on the raw data will be implemented until the main results are published in an open-access journal.

REFERENCES:
- [Background] Campos L, Dias P, Costa M, Rabin L, Miles R, Lestari S, Feraihan R, Pant N, Sriwichai N, Boonchieng W, Yu L. Mental health literacy questionnaire-short version for adults (MHLq-SVa): validation study in China, India, Indonesia, Portugal, Thailand, and the United States. BMC Psychiatry. 2022 Nov 16;22(1):713. doi: 10.1186/s12888-022-04308-0. PMID 36384505
- [Background] INCB. (n.d.). Report of the International Narcotics Control Board for 2021.
- [Background] World Health Organization - Regional Office for Europe. (2015). The European Mental Health Action Plan 2013-2020. World Health Organization, 19.
- [Background] Roth GA, Mensah GA, Johnson CO, Addolorato G, Ammirati E, Baddour LM, Barengo NC, Beaton AZ, Benjamin EJ, Benziger CP, Bonny A, Brauer M, Brodmann M, Cahill TJ, Carapetis J, Catapano AL, Chugh SS, Cooper LT, Coresh J, Criqui M, DeCleene N, Eagle KA, Emmons-Bell S, Feigin VL, Fernandez-Sola J, Fowkes G, Gakidou E, Grundy SM, He FJ, Howard G, Hu F, Inker L, Karthikeyan G, Kassebaum N, Koroshetz W, Lavie C, Lloyd-Jones D, Lu HS, Mirijello A, Temesgen AM, Mokdad A, Moran AE, Muntner P, Narula J, Neal B, Ntsekhe M, Moraes de Oliveira G, Otto C, Owolabi M, Pratt M, Rajagopalan S, Reitsma M, Ribeiro ALP, Rigotti N, Rodgers A, Sable C, Shakil S, Sliwa-Hahnle K, Stark B, Sundstrom J, Timpel P, Tleyjeh IM, Valgimigli M, Vos T, Whelton PK, Yacoub M, Zuhlke L, Murray C, Fuster V; GBD-NHLBI-JACC Global Burden of Cardiovascular Diseases Writing Group. Global Burden of Cardiovascular Diseases and Risk Factors, 1990-2019: Update From the GBD 2019 Study. J Am Coll Cardiol. 2020 Dec 22;76(25):2982-3021. doi: 10.1016/j.jacc.2020.11.010. PMID 33309175
- [Background] Selim AJ, Rothendler JA, Qian SX, Bailey HM, Kazis LE. The History and Applications of the Veterans RAND 12-Item Health Survey (VR-12). J Ambul Care Manage. 2022 Jul-Sep 01;45(3):161-170. doi: 10.1097/JAC.0000000000000420. PMID 35612387
- [Background] Rosas LG, Rodriguez Espinosa P, Montes Jimenez F, King AC. The Role of Citizen Science in Promoting Health Equity. Annu Rev Public Health. 2022 Apr 5;43:215-234. doi: 10.1146/annurev-publhealth-090419-102856. Epub 2021 Nov 1. PMID 34724389
- [Background] Israel BA, Coombe CM, Cheezum RR, Schulz AJ, McGranaghan RJ, Lichtenstein R, Reyes AG, Clement J, Burris A. Community-based participatory research: a capacity-building approach for policy advocacy aimed at eliminating health disparities. Am J Public Health. 2010 Nov;100(11):2094-102. doi: 10.2105/AJPH.2009.170506. Epub 2010 Sep 23. PMID 20864728
- [Background] Chinn D. Critical health literacy: a review and critical analysis. Soc Sci Med. 2011 Jul;73(1):60-7. doi: 10.1016/j.socscimed.2011.04.004. Epub 2011 May 12. PMID 21640456
- [Background] Villalonga-Olives E, Adams I, Kawachi I. The development of a bridging social capital questionnaire for use in population health research. SSM Popul Health. 2016 Aug 31;2:613-622. doi: 10.1016/j.ssmph.2016.08.008. eCollection 2016 Dec. PMID 29349175
- [Background] Nutbeam, D. (2020). Health literacy as a public health goal: a challenge for contemporary health education and communication strategies into the 21st century. Health Promotion International, 15(3), 259-267.
- See also: Website of the project — https://www.cairproject.eu/